CLINICAL TRIAL: NCT05466357
Title: Department of Neurosurgery, Affiliated Hospital of Nantong University
Brief Title: Application Research on Endoscopic Pseudocapsule-Based Resection for Pituitary Adenomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Subei People's Hospital of Jiangsu Province (Other); The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AREPBRPA
Record Dates: First submitted 2022-05-26; First posted 2022-07-20 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-09

CONDITIONS: Pituitary Adenoma
Keywords: pituitary adenomas; pseudocapsule; the endoscopic endonasal approach
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intracapsular excision of pituitary tumor (Experimental): Literature review was conducted to calculate the excision rate, postoperative recurrence rate and postoperative endocrine improvement of previous endoscopic intracapsular excision of pituitary tumor.
  Interventions: Procedure: Excision of pituitary tumor outside pseudocapsule

INTERVENTIONS:
Procedure: Excision of pituitary tumor outside pseudocapsule — Dedicated high-resolution magnetic resonance imaging (MRI) protocols have been proposed to detect pituitary adenoma and accurately guide surgical removal. To accomplish complete PA removal and minimize the impact on pituitary functions, intraoperative navigation was used to identify the tumor pseudocapsule. Depending on different tumor sizes and pseudocapsule development, investigators adopted different resection strategies. The suspicious tissue was sent to the pathology department for histopathology intraoperatively. Long-term postoperative follow-up imaging and endocrine data were used to evaluate tumor prognosis before and after operation. Standardized management and established biobank is critical for pituitary adenomas.

SUMMARY:
Pituitary adenomas are one of the most common primary central nervous system tumors and have an estimated prevalence of 17%. Management of pituitary adenomas involves a multidisciplinary approach that can incorporate surgical, medical, and/or radiation therapies. Over the last two decades, the endoscopic endonasal approach (EEA) has been extensively developed and refined for the resection of pituitary adenomas (PAs). In recent years, extracapsular resection (ER), which emphasized the importance of the pseudocapsule between the adenoma and surrounding normal gland tissue as a surgical plane, was adopted for more radical resection of the tumor. Therefore, dedicated high-resolution magnetic resonance imaging (MRI) protocols have been proposed to detect pituitary adenoma and accurately guide surgical removal. The evaluation of preoperative imaging for pseudocapsule is very important to the surgical method. Depending on different tumor sizes and pseudocapsule development, investigators adopted different resection strategies. To accomplish complete PA removal and minimize the impact on pituitary functions, intraoperative navigation was used to identify the tumor pseudocapsule, also the suspicious tissue was sent to the pathology department for histopathology intraoperatively. Long-term postoperative follow-up imaging and endocrine data were used to evaluate tumor prognosis. Standardized management and established biobank is critical for pituitary adenomas.

DETAILED DESCRIPTION:
一、Project basis The pseudocapsule was first described by Costello in the early 1900s, which was formed by the compression between the tumor and normal gland. Adenoma growth leads to compression of the acinar structure of the adjacent normal gland, resulting in a reticulin-rich pseudocapsule that encases the entire adenoma in. Over the last two decades, the endoscopic endonasal approach (EEA) has been extensively developed and refined for the resection of pituitary adenomas (PAs). The endoscopic panoramic view is superior in terms of efficacy and safety for sellar surgery, and studies have reported that PAs can be effectively resected by EEA with minimal postoperative morbidity. Oldfield and colleagues used the phrase "surgical capsule of adenoma" to describe the histologically confirmed pseudocapsule in 2006 which was found in about 50% of patients and tends to be more frequent in larger tumors. The studies elaborated procedure along the outer face of the pseudocapsule between the adenoma and surrounding normal gland tissue achieved radical removal of the tumor while preserving normal pituitary function. Thus, in recent years, extracapsular resection (ER), which emphasized the importance of pseudocapsule as a surgical plane, was adopted for more radical resection of the tumor.

In smaller tumors, the pseudocapsule tended to exist more prominently and to cover the whole tumor, whereas in larger tumors the pseudocapsule tended to be discontinuous or disrupted. Similarly, in the present study, investigators found that ER was more performed in microadenomas, whereas intracapsular resection (IR) was more adopted in macroadenomas. Furthermore, in some macroadenomas, the pseudocapsule could not be seen until proper intracapsular debulking. By contrast, some PAs exhibited no or undefinable pseudocapsule; during the entire procedure, the adenoma was excised piecemeal progressively with a dissector, blunt ring curette, and aspirator.

Although PAs were frequently present within the pseudocapsule and complete tumor resection using the ER technique has been reported to maximize the effectiveness for PAs with pseudocapsules, many authors believe that resection without compromising pituitary function is imperative to improving the ultimate health outcome of patients. In some selective cases, an incomplete adenoma resection is advised because it is expected that this is best for the patients, through lower complication rates and preserving pituitary function. The actual effects of ER-based complete resection of PA are still under debate.

Intact pituitary gland function is deemed more important than adenoma total removal, Theoretically, it is hard for surgeons to extirpate only tumor cells completely during surgery without removing any normal pituitary gland tissue because in most cases the adenoma directly contacts with the normal pituitary gland. Some scholars found that the capsule itself contains tumor cells and may be a main cause of persistent hypersecretion of the hormone and possibly the source of recurrence. In addition, some studies found that the pseudocapsule is disrupted by tumor invasion so that the extracapsular removal and management of tumor invasion outside of the pseudocapsule are crucial to accomplishing complete PA removal. For these refractory pituitary adenomas, some research recommend aggressive resection, especially in IR resection cases. Partial gland resection or resection of the cavernous sinus medial wall is necessary in some cases since studies showed that it could help improve biochemical remission for the pituitary gland.

Pseudocapsule-Based Resection for Pituitary Adenomas has become a hot topic in recent years. However, it often focuses on the influence of pituitary function after surgical resection and the management and evaluation of surgical complications. How to strengthen the recognition of normal pituitary and pituitary pseudocapsule by imaging before operation? How to combine preoperative image enhanced recognition of pseudocapsule during operation? How to confirm the boundary between normal tissue and pituitary gland by Intraoperative pathology? What kind of treatment strategy should be adopted for pituitary adenomas of different sizes? There are few relevant reports on the above doubts. Standardized operation for pituitary adenoma is also lack, even if it can reduce trauma and complications; There are few studies on relationship among postoperative magnetic resonance imaging and related endocrine function examination and the evaluation of Extr-apseudocapsular resection for Pituitary Adenomas. It is urgent to establish a biological sample bank of pituitary tumor.

二、Research Contents:

1. To identify the pituitary tissue and the pseudocapsule by preoperative imaging data.
2. To evaluate the significance of preoperative imaging by relationship between tumor and pseudocapsule during operation.
3. To research the significance of intraoperative rapid pathology in excision of pituitary tumor
4. To establish Standardized surgical treatment strategies for pituitary tumors.
5. Postoperative imaging data and clinical endocrine function examination were used to evaluate the surgical efficacy.
6. To establish biological sample bank of pituitary tumor.

三、Research method, technical route and work plan

1. General Data and Clinical Manifestations In this retrospective study, investigators will review patients in our and cooperation institutions (Department of Neurosurgery, Affiliated Hospital of Nantong University, Jiangsu, China; Department of Neurosurgery, Subei People's Hospital of Jiangsu province, China; Department of Neurosurgery, The First People's Hospital of Changzhou, Jiangsu, China) who undergo EEA for PAs. The information will collect from patients' electronic medical records included presenting symptoms, operative notes, postoperative course,, laboratory data. Informed consent will obtain from all patients.
2. Endocrinological Evaluations All patients undergo a baseline preoperative pituitary hormone examination including serum cortisol, free thyroxine, thyroid stimulation hormone (TSH), adrenocorticotropic hormone (ACTH), growth hormone (GH) and insulin-like growth factor-1 (IGF-1), prolactin (PRL), luteinizing hormone (LH) and follicle stimulating hormone (FSH), testosterone (in males), and estradiol (in females). Postoperative biochemical remission will be defined as a nadir serum GH level of 3,000 ml/day. Hormonal status will be evaluated at 1 week and 3 months after surgery and twice per year thereafter to evaluate anterior pituitary functions.
3. Imaging Analysis All patients undergo high-resolution magnetic resonance imaging (MRI) examination before operation, within 3 days, 3 months, 6 months, and twice per year after surgery. The distribution and density of the pituitary gland could be seen on T1-weighted MR images. The position of the anterior communicating artery and internal carotid artery could be seen on T2-weighted images, also enabling us to reduce the surgical risks. Computed tomography is useful for demonstrating the degree of pneumatization and locations of septations in the sphenoid sinus. The degree of resection was calculated by measuring the residual tumor volume using MRI data. The magnetic resonance imaging (MRI) scanning was performed before surgery to provide excellent details about the tumor's size and texture, especially to distinguish the boundary between the location of normal adenohypophysis and pseudocapsule.
4. Pathological Examinations All resected tumor tissues were evaluated by routine pathological and immunohistochemical examination. The composition of complete and fragmentary pseudocapsules was pathologically examined. All tissues obtained in the study were paraformaldehyde fixed and paraffin embedded. The sections were stained using hematoxylin and eosin staining or Masson's trichrome staining.

   Intact pituitary gland function is deemed more important than adenoma total removal, Theoretically, it is hard for surgeons to extirpate only tumor cells completely during surgery without removing any normal pituitary gland tissue because in most cases the adenoma directly contacts with the normal pituitary gland.To minimize the impact on pituitary functions, the suspicious tissue was sent to the pathology department for histopathology intraoperatively.
5. Treatment strategies for different types of pituitary tumors Non-function pituitary adenoma, PRL, GH, ACTH
6. Depending on different tumor sizes and pseudocapsule development, investigators adopted different resection strategies.

In microadenoma, the exposed surface of the pituitary gland looks completely normal; a small cut was made in the gland at the location where the adenoma is expected according to preoperative imaging. The right dissector was used to separate the tumor and to preserve the integrity of the pseudocapsule, and achieved total extracapsular resection. Usually, the microadenoma texture is soft, limiting the option of extracapsular dissection. With small ring curettes, the tumor is removed and the tumor cavity was explored meticulously.

For macroadenomas, no attempt is made to remove the entire tumor or pull it forward during the initial phases of the dissection. After the intracapsular tumor is debulked and partially removed followed by a median-lateral or basal-superior order, the residual tumor was separated carefully along the pseudocapsular interface.

If the pseudocapsule was not visible in the first stage, investigators used conventional conservative intracapsular resection. Internal debulking was continued until visualization of the pseudocapsule or cavernous sinus wall was achieved. Extracapsular resection was continued along the plane, preserving as much integrity of the pseudocapsule as possible.

After internal debulking, if the pseudocapsule was still unidentifiable, the adenoma was excised piecemeal progressively. Noteworthily, investigators adopted intensive excision and meticulous sweeping to remove small remnants that are hidden behind the fibrin membranes for PA. The surface of the pituitary gland was peeled off as thin a slice as possible, and the tumor bed was circumferentially resected to remove any small tumor remnant in Cushing disease or acromegaly patients.

To minimize the impact on pituitary functions, the suspicious tissue was sent to the pathology department for histopathology intraoperatively.

ELIGIBILITY:
Inclusion criteria:

According to guidelines for treatment of pituitary tumors，Patients can be eligible for surgery.

Exclusion criteria:

1. Patients with other primary endocrine diseases.
2. Patients with obviously suprasellar and parasellar extensions or with cavernous sinus invasion (grade 4 of knosp classification ).
3. Patients with recent nasal trauma.
4. Patients with nasal infection or/and sphenoid sinus inflammation.
5. Patients with with abnormal coagulation.
6. Patients with other serious diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence | Change from baseline (before operation), within 3 days, 3 months, 6 months, 1 year and 2 years after surgery
  All patients undergo high-resolution magnetic resonance imaging (MRI) examination before operation, within 3 days, 3 months, 6 months, and twice per year after surgery. The degree of resection was calculated by measuring the residual tumor volume using MRI data. Comparing preoperative and postoperative tumor imaging changes, investigators will assess the helpfulness of preoperative imaging judgments for intraoperative tumor resection, and compare the efficacy of different surgical modalities.
Endocrine change | 24 hours, 1 week, 1 month, 3 months, 6 months and 1 year after surgery
  All patients undergo a baseline preoperative pituitary hormone examination. Hormonal status will be evaluated at 24 hours, 1 week, 1 month and 3 months after surgery and twice per year to evaluate anterior pituitary functions. Comparing preoperative and postoperative endocrine reduction, investigators will assess efficacy among different groups and different types of pituitary tumors.

SECONDARY OUTCOMES:
Including incidence of cerebrospinal fluid leakage | Followed up for 2 weeks
  In this retrospective study, investigators will evaluate patients in our and cooperation institutions (Department of Neurosurgery, Affiliated Hospital of Nantong University, Jiangsu, China; Department of Neurosurgery, Subei People's Hospital of Jiangsu province, China; Department of Neurosurgery, The First People's Hospital of Changzhou, Jiangsu, China) who undergo EEA for PAs. Including incidence of cerebrospinal fluid leakage will collect from patients electronic medical records. Informed consent will obtain from all patients. All these characteristics will be compared with preoperation. Investigators will assess differences among different groups.
Incidence of intracranial infection | Followed up for 2 weeks
  In this retrospective study, investigators will evaluate patients in our and cooperation institutions (Department of Neurosurgery, Affiliated Hospital of Nantong University, Jiangsu, China; Department of Neurosurgery, Subei People's Hospital of Jiangsu province, China; Department of Neurosurgery, The First People's Hospital of Changzhou, Jiangsu, China) who undergo EEA for PAs. Incidence of intracranial infection will collect from patients electronic medical records. Informed consent will obtain from all patients. All these characteristics will be compared with preoperation. Investigators will assess differences among different groups.
Incidence of visual and visual impairment | Followed up for 2 weeks
  In this retrospective study, investigators will evaluate patients in our and cooperation institutions (Department of Neurosurgery, Affiliated Hospital of Nantong University, Jiangsu, China; Department of Neurosurgery, Subei People's Hospital of Jiangsu province, China; Department of Neurosurgery, The First People's Hospital of Changzhou, Jiangsu, China) who undergo EEA for PAs. Incidence of visual and visual impairment will collect from patients electronic medical records（Visual acuity will be measured according to the visual acuity standard comparison table, and the visual field will be operated according to the automatic visual field instrument). Informed consent will obtain from all patients. All these characteristics will be compared with preoperation. Investigators will assess differences among different groups.
Incidence of subthalamic injury | Followed up for 2 weeks
  In this retrospective study, investigators will evaluate patients in our and cooperation institutions (Department of Neurosurgery, Affiliated Hospital of Nantong University, Jiangsu, China; Department of Neurosurgery, Subei People's Hospital of Jiangsu province, China; Department of Neurosurgery, The First People's Hospital of Changzhou, Jiangsu, China) who undergo EEA for PAs. Incidence of subthalamic injury will collect from patients electronic medical records. Informed consent will obtain from all patients. All these characteristics will be compared with preoperation. Investigators will assess differences among different groups.

CONTACTS AND LOCATIONS:
Overall Officials: xiao mingbing, MD, Principal Investigator — Affiliadted hospital of nantong university
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cushing H. III. Partial Hypophysectomy for Acromegaly: With Remarks on the Function of the Hypophysis. Ann Surg. 1909 Dec;50(6):1002-17. doi: 10.1097/00000658-190912000-00003. No abstract available. PMID 17862444
- [Result] Jankowski R, Auque J, Simon C, Marchal JC, Hepner H, Wayoff M. Endoscopic pituitary tumor surgery. Laryngoscope. 1992 Feb;102(2):198-202. doi: 10.1288/00005537-199202000-00016. No abstract available. PMID 1738293
- [Result] Hardy J. Transsphenoidal hypophysectomy. 1971. J Neurosurg. 2007 Aug;107(2):458-71. doi: 10.3171/JNS-07/08/0458. No abstract available. PMID 17695407
- [Result] Costello RT. Subclinical Adenoma of the Pituitary Gland. Am J Pathol. 1936 Mar;12(2):205-216.1. No abstract available. PMID 19970261
- [Result] Oldfield EH, Vortmeyer AO. Development of a histological pseudocapsule and its use as a surgical capsule in the excision of pituitary tumors. J Neurosurg. 2006 Jan;104(1):7-19. doi: 10.3171/jns.2006.104.1.7. PMID 16509142
- [Result] Lee EJ, Ahn JY, Noh T, Kim SH, Kim TS, Kim SH. Tumor tissue identification in the pseudocapsule of pituitary adenoma: should the pseudocapsule be removed for total resection of pituitary adenoma? Neurosurgery. 2009 Mar;64(3 Suppl):ons62-9; discussion ons69-70. doi: 10.1227/01.NEU.0000330406.73157.49. PMID 19240574
- [Result] Taylor DG, Jane JA, Oldfield EH. Resection of pituitary macroadenomas via the pseudocapsule along the posterior tumor margin: a cohort study and technical note. J Neurosurg. 2018 Feb;128(2):422-428. doi: 10.3171/2017.7.JNS171658. Epub 2017 Aug 18. PMID 28820308
- [Result] Nagata Y, Takeuchi K, Yamamoto T, Ishikawa T, Kawabata T, Shimoyama Y, Inoshita N, Wakabayashi T. Peel-off resection of the pituitary gland for functional pituitary adenomas: pathological significance and impact on pituitary function. Pituitary. 2019 Oct;22(5):507-513. doi: 10.1007/s11102-019-00980-w. PMID 31377966
- [Result] Li QX, Wang WH, Wang XX. Various Strategies of Transsphenoidal Pseudocapsule-Based Extracapsular Resection in Noninvasive Functional Pituitary Adenomas and their Effectiveness and Safety. Neurol India. 2019 Nov-Dec;67(6):1448-1455. doi: 10.4103/0028-3886.273628. PMID 31857533